CLINICAL TRIAL: NCT05483530
Title: A Phase 1 Clinical Study to Investigate the Safety, Tolerability and Efficacy of HLX60 (Anti-GARP Monoclonal Antibody) Combination With HLX10 (Anti-PD-1 Monoclonal Antibody) in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Study to Investigate the Safety, Tolerability and Efficacy of HLX60 Combination With HLX10 in Subjects With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX60HLX10-FIH101
Record Dates: First submitted 2022-07-06; First posted 2022-08-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-08

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX60 combined with HLX10 (Experimental)
  Interventions: Biological: HLX60 combined with HLX10

INTERVENTIONS:
Biological: HLX60 combined with HLX10 — five various doses of HLX60 combined with flat dose of HLX10

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of HLX60 combined with HLX10 in order to determine the maximum tolerated dose (MTD) and Recommended Phase 2 dose (RP2D) and to evaluate the preliminary efficacy for each combination regimen.

DETAILED DESCRIPTION:
Accelerated titration and "3 + 3" dose escalation were used in this trial . various doses of HLX60(anti-GARP) combined with HLX10(anti-PD-1) by intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced malignant solid tumor, who have failed or cannot receive the standard treatment;
* With at least one evaluable lesion according to RECIST v1.1 (for solid tumors);
* Patients must be able to supply adequate tumor tissue for biomarker (including the expression of PD-L1, GARP) analyses;
* Life expectancy longer than three months;
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.

Exclusion Criteria:

* Has a concurrently active second malignancy, other than adequately treated non-melanoma skin cancers, in situ melanoma or in situ cervical cancer. Participants with history of the second malignancy have been disease-free for <3 years.
* Has a history of (non-infectious) interstitial lung disease (ILD) that required steroids, currently has ILD, or when suspected ILD cannot be ruled out by imaging at screening.
* Participant has unresolved AEs ≥ Grade 2 from prior anticancer therapy except for alopecia.
* Those who have received anti-GARP or anti-GARP/TGFβ complex antibody therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Through study completion, assessed up to 2 years.
  Incidence and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 for patients receiving study drug.
Incidence of DLT | Up to 3 weeks.
  Ratio of the number of patients with DLT events in each dose group to the number of patients in the dose group during the DLT evaluation period.
MTD | Up to 3 weeks.
  The maximum tolerated dose (MTD) of HLX60 combined with HLX10
RP2D | Through study completion, assessed up to 2 years.
  The recommended phase II dose (RP2D) of HLX60 combined with HLX10

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, assessed up to 2 years.
  Percentage of patients with complete response or partial response determined by investigators according to RECIST v1.1
Progression-free survival (PFS) | Through study completion, assessed up to 2 years.
  PFS is defined as the time from the first administration of HLX60 and HLX10 to the first occurrence of disease progression or death due to any cause, whichever occurs first.
Overall survival(OS) | Through study completion, assessed up to 2 years.
  OS is defined as the time from the first administration of HLX60 to death due to any cause.
Cmax | 1 year
  serum concentration (Cmax)
Tmax | 1 year
  time to reach Cmax (Tmax)
t1/2 | 1 year
  elimination half-life (t1/2)
AUC | 1 year
  area under the serum concentration-time curve (AUC)
PD | 1 year
  include the GARP receptor occupancy on Treg cells, tumor infiltrating lymphocytes (TILs), FOXP3, pSMAD 2/3 in tumor tissues.
immunogenicity of HLX60 | 1 year
  Incidence of HLX60 anti-drug antibody (ADA) and neutralizing antibody (NAb)
Potential prognostic and predictive biomarkers | 1 year
  include the expressions of GARP, PD-L1 in tumor tissues and soluble GARP in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Macquarie University Hospital & Nepean Hospital, Sydney, Australia